CLINICAL TRIAL: NCT05455398
Title: Sun Yat-sen Memorial Hospital, Sun Yat-sen University
Brief Title: Establishment of a Trans-round Window Inner Ear Continuous Drug Delivery System for the Treatment of Severe-to-profound Sudden Sensorineural Hearing Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYS-Q-202106
Record Dates: First submitted 2022-06-26; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Hearing Loss, Sudden
MeSH Terms: conditions — Hearing Loss, Sudden

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Round window niche enlargement group (Experimental): The round window niche was surgically removed by general anesthesia, the round window membrane was opened as entirely as possible, and the blockage of the round window membrane was carefully identified.
  Interventions: Procedure: Surgical treatment of round window niche enlargement via round window for inner ear drug delivery
- Drum chamber injection group (Active Comparator): Methylprednisolone (40 mg) was injected via puncture in the posterior quadrant of the tympanic membrane once daily for 7 d. Patients were instructed to remain supine for 30 min to keep the drug in the tympanic chamber and to avoid swallowing to prevent drug flow from the eustachian tube.
  Interventions: Procedure: Drum chamber drug injection

INTERVENTIONS:
Procedure: Surgical treatment of round window niche enlargement via round window for inner ear drug delivery — The round window niche is surgically removed and the hormone is slowly released into the inner ear using a gelatin sponge that has absorbed the hormone in the round window
  Arms: Round window niche enlargement group
Procedure: Drum chamber drug injection — Injection of drugs into the tympanic chamber through the tympanic membrane
  Arms: Drum chamber injection group

SUMMARY:
The investigators enrolled patients with total sudden deafness who had failed treatment with systemic combined intra-dural hormone injections. The patients were randomly divided into a pilot group and a control group for a randomized controlled clinical study, with the pilot group receiving a round window niche enlargement via round window inner ear administration and the control group receiving regular intra-drum injection hormone therapy

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, ≤ 65 years old
2. The diagnostic criteria for total deafness type of sudden deafness published in 2015 were met, and the patient had sudden, unilateral full-frequency severe or very severe sensorineural deafness with or without deafness, tinnitus, peri-aural numbness, vertigo, and dizziness, and the diagnosis of sudden deafness was supported by physical examination, pure tone audiometry(PTA), acoustic impedance, and auditory brainstem response(ABR). Magnetic resonance(MR) of the internal auditory tract ruled out the occupancy of the internal auditory tract and pontocerebellar region.
3. Those with an onset of ≤ 6 weeks who have received a systemic application of glucocorticoid shock therapy, glucocorticoid intra-drum injections, and medication to improve inner ear circulation, but have not responded to treatment (PTA improvement < 15 dB).
4. No history of middle or inner ear surgery, no history of radiotherapy or chemotherapy; no general anesthesia - contraindication.
5. Patients voluntarily participate in this study and sign an informed consent form

Exclusion Criteria:

1. Bilateral sudden deafness, drug-based deafness, autoimmune diseases, specific infections, syndromic deafness malignant tumors.
2. Pregnant and lactating women.
3. Cannot tolerate general anesthesia surgery, and severe liver and kidney dysfunction.
4. Any other conditions that the investigator believes should be excluded from this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Establishment of a trans-round window inner ear continuous drug delivery system for the treatment of severe-to-profound sudden sensorineural hearing loss | up to one year
  Assessment of post-operative hearing improvement by pure tone audiometry

CONTACTS AND LOCATIONS:
Overall Officials: Zhigang ZHANG, master, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No